CLINICAL TRIAL: NCT07254806
Title: A Prospective, Randomized, Double-Blinded, Sham-Controlled, Multicenter Study to Evaluate the Safety and Efficacy of IDCT in Subjects With Single-Level, Symptomatic Mild to Moderate Lumbar Intervertebral Disc Degeneration
Brief Title: A Study to Evaluate the Effectiveness of IDCT (Intradiscal Cell Therapy) in Subjects With One Level, Symptomatic Mild to Moderate Lumbar Degenerative Disc Disease
Acronym: IDCT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: DiscGenics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DGX-A02
Record Dates: First submitted 2025-11-17; First posted 2025-11-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Degenerative Disc Disease
Keywords: DDD; low back pain; degenerative disc disease
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: All parties in this trial will be blinded with the exception of the unblinded injecting sub-investigator and their team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IDCT (n=108); Intradiscal injection of IDCT in a single target disc (Experimental): 1 mL intradiscal injection of 9,000,000 cells/mL
  Interventions: Biological: IDCT (rebonuputemcel)
- Sham (n=54); (Sham Comparator): Needle insertion up to the annulus of a single target disc.
  Interventions: Other: Sham (No Treatment)

INTERVENTIONS:
Biological: IDCT (rebonuputemcel) — Single intradiscal injection of 1 mL of 9,000,000 cells/mL IDCT in a single target disc.
  Arms: IDCT (n=108); Intradiscal injection of IDCT in a single target disc
Other: Sham (No Treatment) — Single Sham needle insertion up to the annulus of a single target disc.
  Arms: Sham (n=54);

SUMMARY:
This is a Phase III, randomized, double-blinded, Sham-controlled, multi-center study in subjects with single-level, symptomatic lumbar (L3- S1) intervertebral disc degeneration. The study will have a 52-week primary period followed by 52 week Follow-up Period (total of 104 weeks).

The study protocol will be approved by the Institutional Review Board (IRB) or Independent Ethics Committee (IEC), and the study will be conducted in accordance with Good Clinical Practice (GCP). All subjects will provide written informed consent prior to Screening.

Approximately 162 subjects will be enrolled in the study. Up to 45 days prior to treatment, subjects will be screened for study inclusion, which includes obtaining baseline MRI and X-ray imaging. Imaging results for subjects initially eligible for study participation will be sent to a central imaging vendor for review and confirmation of eligibility, including the number of levels with degeneration. Subjects meeting all inclusion/exclusion criteria will be assigned to the corresponding treatment arm group and subsequently randomized to IDCT or Sham.

Randomization will occur approximately 7 to 14 days prior to the scheduled treatment administration date.

Overall, 162 subjects will be enrolled and randomized to IDCT or Sham in a 2:1 ratio.

* IDCT (n=108)
* Sham (n=54)

DETAILED DESCRIPTION:
Adult subjects with a diagnosis of single-level, mild to moderate, symptomatic lumbar (L3-S1) intervertebral disc degeneration that give consent and meet all the inclusion criteria and none of the exclusion criteria will be enrolled in this study. The disease, single-level disc will be known as the 'target disc' and will be either L3/L4, L4/L5, or L5/S1.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of mild to moderate, symptomatic, single-level degenerative disc disease (DDD) from L3-S1.
2. Has a target disc that meets Modified Pfirrmann Grade 3-7.
3. Is ≥18 and ≤75 years of age, skeletally mature, and has a body mass index (BMI) ≥18 kg/m2 and ≤38 kg/m2 at Screening.
4. Has been experiencing chronic low back pain for at least 6 months prior to Screening.
5. Has had low back pain that is unresponsive to at least 3 months of conservative care (nonoperative treatment) to include at least one non-pharmacological intervention which may include physical therapy, acupuncture, chiropractic manipulation, massage, and at home medically supervised exercise program and two pharmacological interventions which may include NSAIDs, acetaminophen, duloxetine, and/or injectable therapy.
6. Has pre-treatment low back pain score of 45 to 90 on VAS (Visual Analogue Scale) for low back pain at Screening and Day 1.
7. Has pre-treatment ODI score of 35 to 90 at Screening and Day 1.
8. Is willing to voluntarily sign the informed consent form and agrees to the release of previous medical history for purposes of this study (i.e., HIPAA authorization) at Screening.
9. Is physically and mentally able to comply with the protocol, able to understand and complete the required forms, and willing and able to adhere to the requirements of the protocol in the opinion of the Investigator.
10. Female-born subjects of childbearing potential must agree to and comply with using highly effective methods of birth control for the duration of the study (e.g., oral contraceptive, implant, injectable, indwelling intrauterine device, sexual abstinence, condoms, or a vasectomized partner).-

    Exclusion Criteria:

    Physical/ Medical History Exclusion Criteria
11. Has low back pain that in the Investigator's opinion is predominately myofascial in nature.
12. Has constant, unchanging low back pain that is not improved in any spinal position.
13. Has radiculopathy resulting from nerve compression.
14. Has non-radicular unilateral or bilateral leg pain with intensity greater than 50% of the intensity of the low-back pain, as measured by VAS.
15. Leg pain that is of radicular origin, i.e., due to stimulation of nerve roots or dorsal root ganglion of a spinal nerve by compressive forces.
16. Has frequent leg pain that extends below the knee.
17. Has severe unilateral or bilateral osteoarthritis of the knee or hip.
18. Severe spinal arthritis
19. Has cauda equina syndrome.
20. Has had previous lumbar spine surgery.
21. Has had previous disc invasive treatment procedures (i.e., intradiscal electrothermal therapy, intradiscal radiofrequency thermocoagulation) or intradiscal injections (i.e., injection of corticosteroids, methylene blue, dextrose, or glucosamine and chondroitin sulfate) or diagnostic discography at L3-S1 within the 3 months prior to Screening.
22. Subjects who have had basivertebral nerve ablation at L3-S1.
23. Has clinical suspicion of facet pain as the primary pain generator.
24. Has current infection at the planned procedure site, active systemic infection, or current or prior history of lumbar spinal infection (i.e., discitis, septic arthritis, epidural abscess).
25. Has a history of fibromyalgia.
26. Has tested positive for Hepatitis B virus (HBV), Hepatitis C virus (HCV), or Human Immunodeficiency Virus (HIV).
27. Has presence of an active malignancy or tumor, or a prior history of malignancy within the last five years (except for basal cell carcinoma of the skin).
28. Has presence or prior history of a spinal malignancy.
29. Has significant systemic disease, such as unstable angina or autoimmune disease, such as rheumatoid arthritis. Has a history of congenital or acquired coagulopathy or thrombocytopenia.

31. Is currently taking anticoagulant, antiplatelet, or thrombolytic medications (except for aspirin or nonsteroidal anti-inflammatory drugs [NSAIDS]) and at the Investigator's medical discernment and discretion is unable to withhold medications for the time required per site standard or care, prior to the IDCT injection or is taking antineoplastic medications.

32. Is at higher risk for post-surgical infection (e.g., taking immunosuppressants), has a severe infection or a history of serious infection.

33. Has concomitant conditions requiring daily oral steroid usage for more than 30 days in the preceding 90 days before Screening.

34. Is taking opioids greater than 20 MME per day on an intermittent (as needed) basis OR is taking 20 MME or greater daily for more than 3 months prior to Screening

35. Has a history of unexplained, easy, or persistent bruising or bleeding, bleeding from the gums, or bleeding problems experienced in previous surgical procedures.

36. Has a history of hypersensitivity or anaphylactic reaction to bovine products, sodium hyaluronate/ hyaluronan/ hyaluronic acid, gentamicin, amphotericin b, dimethyl sulfoxide (DMSO), crustaceous/ shellfish, or porcine products.

37. Has an uncontrolled psychiatric condition or substance/alcohol abuse that would potentially interfere with the subject's participation in the study within 2 years prior to Screening in the opinion of the Investigator.

38. Has positive serum pregnancy test or nursing at time of Screening or has plans to become pregnant within the planned length of the study (2 years).

39. Has a body habitus that precludes adequate fluoroscopic visualization for the procedure or the procedure is physically impossible.

40. Has or requires an implantable electronic defibrillator, pacemaker, or has other contraindication to MRI scanning or cannot tolerate MRI scanning. Subjects who are expected to require a defibrillator or pacemaker, as determined by the Investigator should be excluded.

41. Has participated in another clinical study within the 6 months prior to Screening.

42. Has been a recipient or plans to be a recipient during trial participation of stem cell product to treat the lumbar spine.

43. Has participated in a prior IDCT clinical study.

44. Has pending litigation against a health care professional, except where required by the insurer as a condition of coverage.

45. A person who would not be available for the entire planned length of the trial.

46. Has active or pending worker's compensation claims. 47. In the Investigators opinion, the subject is not suitable for participation in the clinical trial.

Imaging Exclusion Criteria:

48. Two or more discs (L3-S1) that have a Modified Pfirrmann Grade 3-7.

49. Has evidence of prior lumbar vertebral body fracture at L3-S1.

50. Has scoliosis with curvature > 10 degrees.

51. Has congenital spinal irregularities such as segmentation.

52. Has an acute fracture of the spine at the time of enrollment in the study. Clinically compromised vertebral bodies within L3-S1 due to current or past trauma, e.g., sustained pathological fracture or multiple fractures of vertebrae.

53. Has evidence of dynamic instability on lumbar flexion extension per screening radiographs as indicated by >4.5 mm of translational motion at L3-S1; >15° of angular motion at L3/-L4; >20° of angular motion at L4-L/5; or >25° angular motion at L5/-S1.

54. Has Grade 2 or higher spondylolisthesis at L3-S1, as assessed by Meyerding classification.

55. Has lumbar spondylitis or other undifferentiated spondyloarthropathy.

56. Has Modic Type III Changes at L3-S1.

57. Has radiographic evidence or suspicion of a full thickness annular tear at L3-S1.

58. Has evidence of abnormal disc morphology defined as an extrusion or sequestration according to Fardon classification at L3- S1.

59. Has herniation > 3 mm in AP dimension that is associated with nerve root compression.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2027-11-24 (Estimated); Study Completion 2028-11-24 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) for low back pain | Week 52
  VAS is a sliding visual scale of 0 being "no pain" and 100 being "worst pain Imaginable' to assess changesfrom baseline in low back pain compared to Sham
Oswestry Disability Index (ODI) | Week 52
  ODI is a 10-item questionnaire used to measure functional disability in people with low back pain. It is a self-administered tool that assesses how back pain affects daily activities like walking, sleeping, and personal hygiene, with scores ranging from 0% (no disability) to 100% (maximum disability).
Adverse Events | Day 1 to Week 52 in each treatment group.
  Incidence of grade 2 (moderate) or greater AEs and SAEs
Adverse events of special interest | Day 1 to Week 52 in each treatment group
  Incidence of Adverse Events of Special Interest (AESI) to include any symptomatic injury of the target disc including annular tear, disc herniation/extrusion/prolapse as well as discitis.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | Week 4, 12 and 26, 78 and 104
  VAS is a sliding visual scale of 0 being "no pain" and 100 being "worst pain Imaginable' to assess changes from baseline in low back pain
Oswestry Disability Index (ODI) | Week 4, 12 and 26, 78 and 105
  ODI is a 10-item questionnaire used to measure functional disability in people with low back pain. It is a self-administered tool that assesses how back pain affects daily activities like walking, sleeping, and personal hygiene, with scores ranging from 0% (no disability) to 100% (maximum disability).
EQ-5D | Enrollment through Week 104
  EQ-5D is a validated too consisting of a set of questions covering five dimensions, with each dimension having a different severity level.
  1. Mobility: Ranging from "no problems walking about" to "confined to bed". Self-care: Ranging from "no problems with self-care" to "unable to wash or dress myself".
  2. Usual activities: Ranging from "no problems doing my usual activities" to "unable to do my usual activities" (e.g., work, study, housework).
  3. Pain/discomfort: Ranging from "no pain or discomfort" to "extreme pain or discomfort".
  4. Anxiety/depression: Ranging from "not anxious or depressed" to "extremely anxious or depressed".
  5. Visual Analog Scale (EQ VAS): A scale (typically 0-100) where respondents mark their overall health from "worst imaginable" to "best imaginable".
Disc Volume | Day 1 to Week 104
  MRI assessment of Disc Volume though Week 104
Pain Medication Use | Enrollment to Week 104
  Concomitant pain medication use for low back pain related to the target disc
Concomitant Therapy | Enrollment to Week 104
  Concomitant medical therapy for low back pain (physical therapy, acupuncture, chiropractic manipulation, massage, and at-home, medically supervised exercise program etc.) use for low back pain
Treatment Failure Rate | Enrollment to week 104
  Treatment failure rate (defined as an invasive non-surgical or surgical intervention) directly related to the target disc.
Adverse Events | Enrollment to Week 104
  The incidence of grade 2 (moderate) or greater AEs and SAEs
Adverse Events of Special Interest (AESI) | Enrollment to Week 104
  The incidence of Adverse Events of Special Interest (AESI) observed defined as any one of the followings symptomatic injury of the target disc including annular tear, disc, herniation/extrusion/prolapse or any case of discitis.

OTHER OUTCOMES:
MRI Based evaluations | Enrollment through Week 104
  MRI Evaluation of the lumbar spine will be reported as an aggregate in one report to assess of disc height, Modified Pfirrmann grade, Modic changes, annular tears/fissures, endplate integrity, herniation, and any additional noteworthy observations at 12, 26, 52, 78, and 104.
X-ray evaluation of the lumbar spine | Screening through Week 104
  X-ray evaluation of flexion/extension will be assessed and measure in degrees of angles.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Flood, Study Director — DiscGenics, Inc.
Locations (6):
- United States (6):
  - Injury Care Family Care Research, Boise, Idaho
  - Axis Spine Center, Post Falls, Idaho
  - The Orthopedic Center of St. Louis, St Louis, Missouri
  - Wake Research, Wilmington, North Carolina
  - Carolinas Pain Institute/ Center For Clinical Research, Winston-Salem, North Carolina
  - Semmes Murphey Neurological Clinic, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided